CLINICAL TRIAL: NCT00419614
Title: Retrospective Chart Review on the Association of Pancreaticoduodenectomy Without Pancreatic-Gastrointestinal Anastomosis to Perioperative Morbidity and Mortality
Brief Title: Outcome of Pancreatic Stump Closure Following Resection of Tumors of the Head of the Pancreas.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: PancStumpHYMC
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Chart review evaluating outcome of patients in whom following resection of a tumor involving the head of the pancreas no anastomosis of the pancreatic stump was done to the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven carcinoma of the head of pancreas or other periampullary carcinoma treated by pancreaticoduodenectomy.

Exclusion Criteria:

* Patients undergoing pancreaticoduodenectomy for other indications (i.e. trauma)
* Charts not available for review.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Ashkenazi, M.D., Principal Investigator — Hillel Yaffe Medical Center